CLINICAL TRIAL: NCT01135888
Title: Short Term Effects and Risks of Physical Exercise in Subjects With Hypohidrotic Ectodermal Dysplasia (Christ-Siemens-Touraine Syndrome)
Brief Title: Short Term Effects and Risks of Physical Exercise in Subjects With Hypohidrotic Ectodermal Dysplasia
Status: Completed | Type: Observational
Sponsor: University Hospital Erlangen (Other)
Collaborators: Pervormance GmbH (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Holm Schneider, Professor of Pediatrics, University Hospital Erlangen
Other Study IDs: ED09
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: X-Linked Hypohidrotic Ectodermal Dysplasia; Exercise-induced Rise of Body Temperature
Keywords: hypohidrotic ectodermal dysplasia; exertional hyperthermia; cooling device
MeSH Terms: conditions — Ectodermal Dysplasia 1, Anhidrotic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- HED children
- HED adolescents
  Interventions: Device: Skin cooling devices
- Control children
- Control adolescents
  Interventions: Device: Skin cooling devices

INTERVENTIONS:
Device: Skin cooling devices — Cooling vest and cooling bandana
  Other Names: Cooline
  Groups: Control adolescents; HED adolescents

SUMMARY:
Because of their lack of sweat glands individuals with hypohidrotic ectodermal dysplasia (HED) are at particular risk of life-threatening hyperthermia during exercise in a warm environment. In this study, the effects of physical exercise are investigated in boys and male adolescents with X-chromosomally inherited HED as well as age-matched controls, who undergo standardized exertion on a bicycle ergometer at ambient temperatures of 25°C and 30°C. Body core temperature during and after ergometry, heart rate, performance, and serum lactate as a marker of metabolic stress are measured. Subjects with HED are expected to show an endangering rise of body temperature in connection with physical exercise. To clarify, whether novel cooling devices may reduce the likelihood of overheating, the effects of such devices are evaluated at 30°C.

ELIGIBILITY:
Inclusion Criteria:

* for patients: hypohidrotic ectodermal dysplasia caused by EDA gene mutations
* regular fluid intake prior to the investigation
* written informed consent

Exclusion Criteria:

* acute febrile illness
* acute or chronic heart disease
* arterial hypertension
* gastrointestinal disorders
* implantable electronic devices
* MRI investigation scheduled for the 5 days subsequent to the study
* clinical signs or diagnostic findings of dehydration

Ages: 7 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: subjects with X-chromosomally inherited hypohidrotic ectodermal dysplasia (HED) and age-matched controls
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holm Schneider, MD, Principal Investigator — University Hospital Erlangen
Locations (1):
- University Hospital Erlangen, Erlangen, Bavaria, Germany

REFERENCES:
- [Derived] Hammersen JE, Neukam V, Nusken KD, Schneider H. Systematic evaluation of exertional hyperthermia in children and adolescents with hypohidrotic ectodermal dysplasia: an observational study. Pediatr Res. 2011 Sep;70(3):297-301. doi: 10.1203/PDR.0b013e318227503b. PMID 21646941